CLINICAL TRIAL: NCT03874377
Title: Examining the Feasibility of a Brief Adjunctive Mindfulness Intervention for Adolescents With Obesity
Brief Title: Mindfulness in Adolescents With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Elizabeth Cotter, Assistant Professor, American University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNMC Pro00011128
Record Dates: First submitted 2019-03-07; First posted 2019-03-14 (Actual); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Mindfulness; Usual Care
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness (Experimental): The mindfulness intervention consists of 6 weekly sessions, blending material from the evidence-based Learning to BREATHE and Mindfulness-Based Eating Awareness Training manualized interventions. Sessions will focus on: experiential mindfulness exercises, such as mindful eating, loving kindness practices, breath awareness, and mindful movement; hunger and satiety awareness; improving responses to emotions; practicing acceptance and being non-judgmental; and tolerating negative feelings and sensations, including those related to hunger and cravings. Participants will be assigned brief homework exercises (approximately 10 minutes) daily in between appointments.Participants in this arm will also receive the usual care provided by the weight management clinic.
  Interventions: Behavioral: Mindfulness; Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness refers to the experience of paying attention to the present moment in a nonjudgmental manner. The mindfulness intervention consists of 6 weekly sessions focused on: experiential mindfulness exercises, such as mindful eating, loving kindness practices, breath awareness, and mindful movement; hunger and satiety awareness; improving responses to emotions; practicing acceptance and being non-judgmental; and tolerating negative feelings and sensations, including those related to hunger and cravings. Participants will be assigned brief homework exercises (approximately 10 minutes) daily in between appointments.
Behavioral: Usual Care — Participants will receive the recommended standard of medical management of overweight and obesity. The clinic team conducts a comprehensive evaluation of the patient to assess dietary and activity behavior change needs of each patient and family, as well as obesity-associated comorbidities. In addition to management of comorbidities, goals for improved physical activity and dietary behaviors are set with the patient and family at each visit.

SUMMARY:
The goal of this study is to conduct a single arm open trial to examine the feasibility of a brief, adjunctive mindfulness intervention tailored to the needs of adolescents with severe obesity.

DETAILED DESCRIPTION:
The purpose of this study is to examine whether it is feasible to integrate a brief, adjunctive mindfulness intervention with the standard medical management of obesity in adolescents with severe obesity. Mindfulness refers to the experience of paying attention to the present moment in a nonjudgmental manner. Mindfulness training enhances one's ability to cope with negative emotions and one's awareness of decision-making processes and internal experiences.

The proposed study has two specific aims: 1) to conduct a single arm open trial to examine the feasibility and acceptability of the mindfulness intervention in a sample of 15 adolescents with severe obesity; and 2) to examine the preliminary efficacy of the mindfulness intervention on BMI, emotion regulation, eating and weight-related behaviors, impulsivity, waist circumference, and blood pressure in comparison to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 12 - 17 years
* a current patient of our affiliated obesity clinic
* have a body mass index (BMI) between 30 and 45 kg/m2.

Exclusion Criteria:

* have a known genetic cause of obesity
* have been diagnosed with a severe intellectual or learning disability
* have been diagnosed with an autism spectrum disorder or current psychosis
* are taking a medication intended to reduce body weight

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Medical Center - IDEAL Clinic, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cotter EW, Hornack SE, Fotang JP, Pettit E, Mirza NM. A pilot open-label feasibility trial examining an adjunctive mindfulness intervention for adolescents with obesity. Pilot Feasibility Stud. 2020 Jun 6;6:79. doi: 10.1186/s40814-020-00621-1. eCollection 2020. PMID 32518670

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness
Started | 11
Completed | 8
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Mindfulness
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.36 (1.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 2
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Sessions Attended by Participant
Description: Retention will be tracked via attendance; research staff will take attendance during each assessment period and intervention session to determine the feasibility of retaining participants.
Time Frame: 6 weeks post study start date
Measure: Number; unit: percentage of all sessions attended
Arm/Group | Mindfulness
Number analyzed (Participants) | 11
percentage of all sessions attended | 85

2. Primary Outcome: Participant Satisfaction: Satisfaction Survey
Description: We will assess participants' satisfaction with the intervention by having them complete a satisfaction survey at the end of the program to assess perceived helpfulness of the intervention and to elicit feedback on the various components. Participants respond to 6 questions (e.g., "I enjoyed being a part of this program") on a scale of 1 (strongly disagree) to 5 (strongly agree). An average across scores will be calculated with higher scores reflecting greater satisfaction. Possible scores range from 1 to 5.
Time Frame: 6 weeks post study start date
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness
Number analyzed (Participants) | 8
score on a scale | 4.5 (.53)

3. Secondary Outcome: Binge Eating - Eating Disorders Examination-Questionnaire (EDEQ).
Description: Participants will report instances of binge eating via items of the Eating Disorders Examination-Questionnaire (EDEQ). Participants report how often they engaged in binge eating over the past 28 days 0 (no days) to 28 (every day). Higher scores represent greater eating pathology.
Time Frame: Change from Baseline to 6 weeks
Measure: Mean (95% Confidence Interval); unit: Number of days
Arm/Group | Mindfulness
Number analyzed (Participants) | 11
Number of days | 3.75 [-3.46 to 10.96]

4. Secondary Outcome: Mindful Attention Awareness Scale-Adolescent (MAAS-A)
Description: Participants rate how frequently they experience episodes of mindless behavior via the Mindful Attention Awareness Scale-Adolescent (MAAS-A). The MAAS-A is a 15-item measure of dispositional mindfulness. Participants respond to statements on a scale from 1 (almost always) to 6 (almost never). Items are summed with scores ranging from 15 to 90, with higher scores representing higher levels of mindfulness.
Time Frame: Change from Baseline to 6 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mindfulness
Number analyzed (Participants) | 11
score on a scale | .20 [-.73 to .32]

5. Secondary Outcome: "Go" Reaction Time - Measure of Inhibitory Control
Description: The Go No Go Task examines inhibitory control via a computerized program. Participants are instructed to press a button when a certain image is shown on the screen (e.g., a green rectangle, a cross). They are instructed not to respond when another image is shown on the screen (e.g., a blue rectangle, an X). Poor inhibitory control is evident by more failures to inhibit responses in the "no go" condition. Reaction time is the processing speed for correct Go trials.
Time Frame: Change from Baseline to 6 weeks
Measure: Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Mindfulness
Number analyzed (Participants) | 11
milliseconds | 34.87 [4.99 to 64.76]

6. Secondary Outcome: Body Mass Index (BMI)
Description: Height and weight will be assessed in order to calculate BMI.
Time Frame: Change from Baseline to 6 weeks
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Mindfulness
Number analyzed (Participants) | 11
kg/m^2 | 2.91 [-3.38 to 9.2]

7. Secondary Outcome: Overeating - Eating Disorders Examination-Questionnaire (EDEQ).
Description: Participants report instances of overeating via items of the Eating Disorders Examination-Questionnaire (EDEQ). Participants report how often they engaged in overeating over the past 28 days 0 (no days) to 28 (every day). Higher scores represent greater overeating.
Time Frame: Change from Baseline to 6 weeks
Measure: Mean (95% Confidence Interval); unit: Number of days
Arm/Group | Mindfulness
Number analyzed (Participants) | 11
Number of days | 1.83 [-.22 to 3.89]

8. Secondary Outcome: Go No Go False Alarm Rate - Measure of Inhibitory Control
Description: The Go No Go Task examines inhibitory control via a computerized program. Participants are instructed to press a button when a certain image is shown on the screen (e.g., a green rectangle, a cross). They are instructed not to respond when another image is shown on the screen (e.g., a blue rectangle, an X). Poor inhibitory control is evident by more failures to inhibit responses in the "no go" condition. The false alarm rate refers to incorrect No Go trials.
Time Frame: Change from Baseline to 6 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of "no gos that are incorrect
Arm/Group | Mindfulness
Number analyzed (Participants) | 11
percentage of "no gos that are incorrect | .06 [-.04 to .17]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Mindfulness
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT03874377/Prot_SAP_000.pdf